CLINICAL TRIAL: NCT04350983
Title: Physical Activity on Prescription and Enhanced Individual Support by Physiotherapist A Comparative Study Between Individuals With One Diagnosis and Multimorbidity
Brief Title: Physical Activity on Prescription and Enhanced Individual Support by Physiotherapist
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Elin Laurila, Physiotherapist, Vastra Gotaland Region
Other Study IDs: PAP enhanced support 271821
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Physical Activity; Sedentary Behavior; Multimorbidity
Keywords: Physical activity on prescription; Individual support; Enhanced support; Person-centered care; Physiotherapist
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Increased physical activity — PAP and enhanced individual support by physiotherapist to increase physical activity

SUMMARY:
Multimorbidity is common, especially in the elderly population and is associated with a higher risk of mortality and disability, lower quality of life, polypharmacy, increased healthcare use and costs. Physical inactivity increases the risk of multimorbidity and individuals with multimorbidity are more likely to be physically inactive. Physical activity can prevent and treat several diseases. Physical Activity on Prescription (PAP) is an evidence-based method used in health care to increase physical activity. The aim of this study was to investigate whether self-reported physical activity level increase and sedentary time decreases in individuals who have received PAP in health care completed with enhanced individual support by physiotherapist at PAP-reception in wellness center for six months and to compare individuals with one diagnosis to individuals with multimorbidity.

The study population consisted of 331 adults who received PAP in health care and enhanced individual support by a physiotherapist at PAP-reception during six months. Data has been collected retrospectively from a local register with questionnaires from the PAP-reception. Self reported physical activity minutes/week and hours of sedentary time/day were measured at baseline and at six months. Differences in physical activity minutes and sedentary time from baseline to six months have been compared between individuals with one diagnosis and individuals with multimorbidity.

ELIGIBILITY:
Inclusion Criteria:

* Received physical activity on prescription from health care
* Contact with PAP-reception

Exclusion Criteria:

Ages: 20 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of men and women aged 20-93 years who received PAP from health care and enhanced individual support by physiotherapist at PAP-reception in wellness centre in central and western Gothenburg in 2015-2016. The majority of the study population had a multimorbidity and the most common diagnosis was musculoskeletal disease.
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Physical activity minutes/week | Change between baseline and six months follow up.
  Self-assessment of two physical activity questions
Sedentary time hours/day | Change between baseline and six months follow up.
  Self-assessment of one sedentary behaviour question

SECONDARY OUTCOMES:
Diagnoses | Measured at baseline
  Type and number of diagnoses
Visits and telephone contacts | Measured at six months follow up
  Number of visits and telephone contacts
Socia demographic data | Measured at baseline
  Age (years), sex (female/male)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Larsson, PhD, Principal Investigator — Sahlgrenska academy, University of Gothenburg

IPD SHARING:
Plan to Share IPD: Yes
The data that supports the findings of this study are available from the corresponding author on reasonable request.